CLINICAL TRIAL: NCT02246140
Title: Prevalence of Intracranial Arterial Stenosis in Regular Resin of Cannabis Users Compared to Control Subjects: a Preliminary Study of Feasibility
Brief Title: Intracranial Arterial Stenosis and Resin of Cannabis Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5715
Record Dates: First submitted 2014-09-17; First posted 2014-09-22 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cannabis Users
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cannabis users (Experimental): Cerebral MRI and MRA
  Interventions: Other: Cerebral MRI and MRA
- healthy volunteers (Active Comparator): Cerebral MRI and MRA
  Interventions: Other: Cerebral MRI and MRA

INTERVENTIONS:
Other: Cerebral MRI and MRA

SUMMARY:
There is an association between intracranial arterial stenosis and ischemic stroke in young adults. The aim of this study is to evaluate the prevalence of intracranial arterial stenosis in asymptomatic regular resin of cannabis users in comparison with control subjects.

ELIGIBILITY:
Inclusion Criteria:

* regular resin of cannabis users

Exclusion Criteria:

* taking vasoactive medications
* taking other illicit drugs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Presence of intracranial arterial stenosis on cerebral MRA | 3 months
  Rate on cerebral MRA the presence of cerebral Intracranial Arterial Stenosis segmental narrowing defined by at least two intra-cranial arteries compared with a cohort of non cannabis controls subjects.

SECONDARY OUTCOMES:
-Silent ischemic stroke on cerebral MRI | 3 months
  Evaluate on cerebral MRI the presence of sequelae of ischemic stroke defined by a parenchymal hyperintensity in a vascular territory defined on a T2 sequence.
-new intracranial arterial stenosis at 3 month follow-up | 3 months
  Evaluate a cerebral MRA at 3 months the presence of new intracranial stenosis among cannabis users, according to the prosecution or stopping use
-Reversibility of intracranial arterial stenosis at 3 month follow-up | 3 months
  Evaluate on cerebral MRA at 3 months reversibility stenosis present at T0 in cannabis users having stopped their consumption

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Wolff, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France